CLINICAL TRIAL: NCT02397382
Title: A Phase 1, Open-label, Drug Interaction Study to Evaluate the Effect of Guselkumab (CNTO 1959) on Cytochrome P450 Enzyme Activities Following a Single Subcutaneous Administration in Subjects With Moderate to Severe Plaque-type Psoriasis
Brief Title: Pharmacokinetic Study to Evaluate the Effect of a Single Dose of Guselkumab (CNTO 1959) on CYP 450 Enzyme Activities After Subcutaneous Administration in Participants With Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR106796; CNTO1959PSO1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Psoriasis
Keywords: Psoriasis; Guselkumab; Cytochromes P450
MeSH Terms: conditions — Psoriasis | interventions — guselkumab; Midazolam; Warfarin; Omeprazole; Dextromethorphan; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Guselkumab and Cytochrome P450 Probe Cocktail (Experimental): Participants will be administered single dose of Guselkumab 200 milligram (mg) by subcutaneous injection (2*100 mg) on Day 8 and Cytochrome P450 probe cocktail consist of midazolam, warfarin/vitamin K, omeprazole, dextromethorphan and caffeine orally once on Day 1,15 and 36.
  Interventions: Drug: Guselkumab; Drug: Midazolam; Drug: Warfarin; Drug: Omeprazole; Drug: Dextromethorphan; Drug: Caffeine

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered as a single dose of 200 milligram (mg) by subcutaneous injection (2*100 mg) on Day 8.
Drug: Midazolam — Midazolam will be administered orally as probe cocktail containing 0.03 mg per kilogram (kg) once on Day 1, 15 and 36.
Drug: Warfarin — Warfarin will be administered orally as probe cocktail containing 10 mg once on Day 1, 15 and 36.
Drug: Omeprazole — Omeprazole will be administered orally as probe cocktail containing 20 mg once on Day 1, 15 and 36.
Drug: Dextromethorphan — Dextromethorphan will be administered orally as probe cocktail containing 30 mg once on Day 1, 15 and 36.
Drug: Caffeine — Caffeine will be administered orally as probe cocktail containing 100 mg once on Day 1, 15 and 36.

SUMMARY:
The purpose of this study is to evaluate the potential effects of a single dose of 200 milligram (mg) guselkumab on the plasma concentrations of a cocktail of representative probe substrates of Cytochrome P450 isozymes (CYP3A4, CYP2C9, CYP2C19, CYP2D6, and CYP1A2) in participants with moderate to severe psoriasis.

DETAILED DESCRIPTION:
This is an open-label, multi-center study. The total duration of study will be approximately 17 weeks per participant, including Screening phase (up to 4 weeks prior to first probe cocktail administration). Participants will have 4 in-patient periods on Day 1, 8, 15 and 36 (3 periods consisting of 3 days and 2 nights each and 1 consisting of 2 days and 1 night) followed by follow up period (up to Day 92). All Participants will receive a single 200 mg subcutaneous (SC) injection (2*100 mg) of guselkumab on Day 8 and probe cocktail on Days 1, 15 and 36. Blood samples will be collected for the evaluation of pharmacokinetics and immunogenicity at pre-dose and post-dose of study treatment. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque-type psoriasis with or without psoriatic arthritis (PsA) for at least 6 months before Day 1
* Have a Psoriasis Area and Severity Index (PASI) greater than or equal to (>=) 12 at Screening
* Have an Investigator's Global Assessment (IGA) >= 3 at Screening
* Have an involved body surface area (BSA) >= 10 percent (%) at Screening
* Be a candidate for phototherapy or systemic treatment for psoriasis

Exclusion Criteria:

* Has a history of or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, cardiac (including unstable cardiovascular disease, defined as a recent clinical deterioration (example, unstable angina, rapid atrial fibrillation) in the last 3 months or a cardiac hospitalization within the last 3 months), vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, bleeding disorder, rheumatologic, psychiatric, or metabolic disturbances
* Have a pulse oximetry value less than (<) 94 % at Screening
* Genetically determined poor metabolizers of CYP2C9, CYP2C19, and CYP2D6 substrates
* Is currently undergoing or has previously undergone allergy immunotherapy for a history of anaphylactic reactions
* Has a transplanted organ (with exception of a corneal transplant greater than (>) 3 months before Day 1)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Screening up to 96 hours on Day 1, 15 and 36
  The Cmax is the maximum observed plasma concentration of Midazolam, Omeprazole, Dextromethorphan, Caffeine and S-warfarin.
Time to Reach Maximum Concentration (Tmax) | Screening up to 96 hours on Day 1, 15 and 36
  The Tmax is time to reach the maximum observed plasma concentration of Midazolam, Omeprazole, Dextromethorphan, Caffeine and S-warfarin.
Area Under the Plasma Concentration-time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Screening up to 96 hours on Day 1, 15 and 36
  The AUC (0-last) is area under the plasma concentration-time curve from time zero to time of last quantifiable concentration of Midazolam, Omeprazole, Dextromethorphan, Caffeine and S-warfarin.
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0 - infinity]) | Screening up to 96 hours on Day 1, 15 and 36
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to extrapolated infinite time.
Serum Concentration of Guselkumab | Pre-dose on Day 8 and up to Day 92
  The observed serum concentration of Guselkumab.
Number of Participants with antibody to CNTO1959 | Pre-dose on Day 8 and up to Day 92
  The frequency of anti-CNTO1959 antibodies.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 92 Days
  The incidence of TEAEs and SAEs from the screening visit and until the follow-up contact will be will be summarized by treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- United States (8):
  - Anniston, Alabama
  - North Hollywood, California
  - Orlando, Florida
  - Atlanta, Georgia
  - High Point, North Carolina
  - Duncansville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - San Antonio, Texas

REFERENCES:
- [Derived] Zhu Y, Xu Y, Zhuang Y, Piantone A, Shu C, Chen D, Zhou H, Xu Z, Sharma A. Evaluating Potential Disease-Mediated Protein-Drug Interactions in Patients With Moderate-to-Severe Plaque Psoriasis Receiving Subcutaneous Guselkumab. Clin Transl Sci. 2020 Nov;13(6):1217-1226. doi: 10.1111/cts.12807. Epub 2020 May 28. PMID 32407591
- See also: A Phase I, Open-label, Drug Interaction Study to Evaluate the Effect of Guselkumab (CNTO 1959) on Cytochrome P450 Enzyme Activities Following a Single Subcutaneous Administration in Subjects with Moderate to Severe Plaque-type Psoriasis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=9675&filename=CR106796_CSR.pdf